CLINICAL TRIAL: NCT07378813
Title: Comparison of Changes in Neuromuscular and Functional Performance Due to Resistance Training With Low-Load or High-Load in Persons With Parkinson's Disease.
Brief Title: Low Versus High Load Training and Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251268
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Activity, Motor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Load Resistance Training (Active Comparator): Participants will receive low-load resistance training, twice per week for at least 24 sessions for up to 12 weeks.
  Interventions: Behavioral: Low-Load Resistance Training
- High-Load Resistance Training (Active Comparator): Participants will receive high-load resistance training, twice per week for at least 24 sessions for up to 12 weeks.
  Interventions: Behavioral: High-Load Resistance Training

INTERVENTIONS:
Behavioral: Low-Load Resistance Training — Participants will receive a total of twenty-four 45-minutes in-person training sessions, twice per week using three sets of eight repetitions per set. During training participants will be allowed 2-minute rests between sets. Exercises will include four upper-body exercises and two lower-body exercises.
  Arms: Low-Load Resistance Training
Behavioral: High-Load Resistance Training — Participants will receive a total of twenty-four 45-minutes in-person training sessions, twice per week using four sets of eight repetitions per set. During training participants will be allowed 2-minute rests between sets. Exercises will include four upper-body exercises and two lower-body exercises.
  Arms: High-Load Resistance Training

SUMMARY:
This study will compare the effects of high-load resistance training to low-load resistance training, on measures of muscle strength and power and tests of daily performance in older adults with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease Hoehn & Yahr Stages 1-3
* Able to walk 50m unassisted
* Able to understand and communicate in English
* A Montreal Cognitive Assessment (MoCA) score above 18

Exclusion Criteria:

* Uncontrolled cardiovascular or other neuromuscular disease that prevent participation in a training program
* Any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, or other serious concomitant medical illness
* Unresolved injury or surgery to the upper or lower limbs that prevents weight training.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in neuromuscular performance as measured by 1-repetition maximum (1RM) | [Time Frame: Baseline, 12 weeks]
  Maximal load that can be lifted in one repetition (1RM) will be assessed in both leg press and chest press exercises. The loads on the testing equipment will be increased across 5 to 7 testing repetitions. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test. The higher the 1RM the stronger the person is. The unit of measurement is kilograms.
Change in neuromuscular performance as measured by Power Production | Baseline, 12 weeks
  This test measures the power a person can produce at maximal speed using loads of 20%, 40%, 60%, 80%, and 90% of 1RM for the chest press and leg press. Power shows how fast a person can do work. Unit of measure is Watts.

SECONDARY OUTCOMES:
Change in the Speed of the Ten-Meter Walk Test. | Baseline, 12 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk at usual walking speed and as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when the 10-m mark is crossed. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed at each speed, and the average will be documented in meters per second. One-minute recoveries will be provided between trials.
Change in Time for the Five Times Sit-to-Stand Test. | Baseline, 12 weeks
  The five-time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with arms folded across the chest and the back against the chair. On a verbal command, the participant will stand up and sit down five times as quickly as possible. Timing begins at the word go and ends when the buttocks touch the chair after the fifth repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Change in the time required to complete the timed Up-and-Go Test. | Baseline, 12 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair and then returns to a seated position as quickly as possible. Time is measured in seconds.
Change in Distance of the Seated Medicine Ball Throw. | Baseline, 12 weeks
  For the Seated Medicine Ball Throw, subjects will sit in an armless chair with the back against the chair back, while holding the 6-pound medicine ball against the chest.
  Subjects will then throw the ball at a perceived 45° angle as far as possible. Subjects must complete at least three practice trials; however, subjects will be allowed more trials until comfortable with the testing procedure. Upon starting the official trial, subjects will complete three separate attempts at each varying medicine ball, to nine trials in total.
  Each of the three trials within a given medicine ball test will be separated by a 1-minute rest. Distance will be measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No